CLINICAL TRIAL: NCT05672394
Title: Efficacy of Perioperative US-Guided Serratus Anterior Plane Block Versus Thoracic Epidural in Adult Patient Undergoing Thoracotomy: A Randomized Comparative Double-Blinded Trial
Brief Title: US-Guided Serratus Anterior Plane Block Versus Thoracic Epidural in Patients Undergoing Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ms-322-2021
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer; Acute Pain; Chronic Pain
Keywords: Lung Cancer; Serratus anterior plane block; Thoracic epidural
MeSH Terms: conditions — Lung Neoplasms; Acute Pain; Chronic Pain | interventions — Tea; Bupivacaine; Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus anterior plane block: (Experimental)
  Interventions: Procedure: Continuous Serratus anterior plane block; Drug: Bupivacaine
- Thoracic Epidural (Active Comparator)
  Interventions: Procedure: Thoracic Epidural; Drug: Bupivacaine; Drug: lidocaine with epinephrine

INTERVENTIONS:
Procedure: Continuous Serratus anterior plane block — in lateral position a linear transducer (10-12MHz, M-Turbo) will be used, The 5th rib is identified in the mid-axillary line. The following muscles are overlying the rib latissimusdorsi ,teres major, and serratus muscle.The needle (22G, 50-mm Tuohy needle) is introduced in-plane targeting the plane superficial to serratus muscle. local anesthetic is injected then a catheter is threaded and . Ultrasound-guided SAPB was done using a serratus anterior catheter Group DL (n=20) received a bolus of 30 mL of 0.25% bupivacaine followed by a continuous infusion of 0.125% bupivacaine at a rate of 7-12 ml/hr according to patient response upon ICU arrival after the stabilization of the clinical status. The infusion was continued until the end of the 1st 24 hours postoperatively .
  Arms: Serratus anterior plane block:
Procedure: Thoracic Epidural — A thoracic epidural catheter was done to the patient while sitting. Tuohy needles are used. Epidural space can be identified by loss of resistance. Injection begins with a negative aspiration and a test dose (3 ccs of 1.5% lidocaine with 1:200,000 epinephrine) .A Continuous epidural technique through the placement of a catheter 3-5 cm beyond the needle is applied. Injection in 5ml increments of 0.25% bupivacaine is used until the block of the required segments achieved ( 10 to 15ml). sensory testing is via pinprick and cold test to detect sympathetic block . Throughout the technique hourly injection of 5 ml 0.25% bupivacaine for maintenance.
  Arms: Thoracic Epidural
Drug: Bupivacaine — bupivacaine
Drug: lidocaine with epinephrine — 3 ccs of 1.5% lidocaine with 1:200,000 epinephrine
  Arms: Thoracic Epidural

SUMMARY:
Thoracic surgeries is known to be one of the most painful surgeries . Multiple analgesic techniques have been used for post operative analgesia including Thoracic epidural , Patient Controlled Analgesia and systemic opioids. Opioids are associated with multiple sied effects including : PONV , Respiratory depression and ileus while thoracic epidural has its own complications such as hemodynamic instability , injury of spinal cord, pneumothorax and epidural hematoma.

Peripheral nerve blocks provide good alternative for perioperative analgesia. The purpose of our study is to compare the effectiveness of perioperative continuous serratus anterior plane block versus continuous thoracic epidural in pain management during thoracic surgeries for malignancy resection.

DETAILED DESCRIPTION:
Thoracic surgeries is known to be one of the most painful surgeries and it is considered the major factor to the morbidity and mortality postoperatively. A variety of analgesic techniques for example; systemic opioid, intercostal nerve blockade, intra-pleural analgesia, an epidural opioid with or without local anesthetic, and patient-controlled analgesia (PCA) via systemic or epidural route has been used very commonly for thoracotomy pain management.The use of systemic opioids alone was associated with a 23.4% incidence of post-thoracotomy pain syndrome. Also, high doses of opioids represent a safety concern due to respiratory depression. The high incidence of postoperative nausea and vomiting (PONV) exacerbates patients' discomfort. Long-acting opioids hinder faster recovery, thereby delaying discharge. , Serratus anterior plane block (SAPB) has been recently introduced as a promising method that can be used between T2 and T9 levels for analgesia in thoracic surgery. SAPB seems to provide its effect through blockade of the lateral cutaneous branches of the intercostal nerves. Previous reports showed that after superficial SAPB the duration of sensory block was between 7 and 12 hrs. Continuous SAPB could represent an important analgesic alternative in patients who have contraindications to thoracic epidural for example patients with coagulopathies. Hence it is important to thoroughly study this block as an analgesic modality in thoracotomies. Moreover, episodes of hypotension during thoracotomies as during vascular clamping are challenging in the presence of thoracic epidural.

The purpose of our study is to compare the effectiveness of perioperative continuous serratus anterior plane block versus continuous thoracic epidural in pain management during thoracic surgeries for malignancy resection. To the best of our knowledge controlled randomized, prospective studies about the use of this technique in thoracotomies for resection of malignancies are lacking and none has been published to discuss this issue. Also, studies reporting patients' satisfaction are lacking.

Aim of the work

This study aims at evaluating the efficacy of applying continuous serratus anterior plane block (SAPB)as a perioperative analgesic modality for thoracic cancer surgeries (mesothelioma and bronchogenic carcinoma) as compared to continuous thoracic epidural as reflected on decreasing perioperative opioids consumption and postoperative VAS.

Hypothesis

We hypothesize that continuous Serratus anterior plane block via an indwelling catheter is effective in the management of pain in thoracic cancer surgeries when compared to thoracic epidural. Continuous SAPB could reduce both intraoperative and postoperative opioid requirements and improve postoperative VAS scores better than or equivalent to thoracic epidural. It may also delay the time to first required analgesic dose. In addition to providing more stable intraoperative hemodynamics. We planned for this study to evaluate this block continuous (SAPB) which can have a positive effect on pain control, ICU stay.

Ethical Considerations This study will be conducted after the approval of the research committee of the department of anesthesia, surgical ICU, and pain management in KasrAlainy Hospital, Cairo University, and the ethical committee of the Faculty of Medicine, Cairo University. Informed consent will be taken from all patients included in the study.

Methodology

* Study design A controlled randomized double blinded comparative study.
* Study setting and location National Cancer Institute - Cairo University

Randomization The participants in this study will be randomized into two groups based on computer-generated numbers using an online randomization program (research randomizer).

Study Protocol The study will include74 patients. 37patients in each group .Preoperative assessment is conducted on the patients that will be enrolled in this study including history taking, physical examination, and routine laboratory investigations; in the form of CBC, coagulation profile, creatinine, urea, ALT, AST, and radiological investigations; according to the medical condition of the patients. All patients should fulfill the inclusion criteria. A written informed consent form will be obtained from the patients that will be enrolled in the study.

Preoperative On the day of surgery, the patient ID will be confirmed in the preparation room, then 22G cannula will be inserted to the patient, premeditations will be given including lactated ringer solution 500ml, midazolam 2mg, ranitidine 50mg & metoclopramide 10mg. VAS scale will be explained to all patients. The patient marks on the line the point that they feel represents their perception of their current state.

Intraoperative: Before induction of anesthesia The patient is allocated in one of 2 groups , This is known to the anesthesiologist inserting the catheter .

Group 1: Serratus anterior plane block:

Patients are placed in the lateral position with the diseased side up. A linear ultrasound transducer (10-12MHz, M-Turbo Ultrasound, USA) is placed over the midclavicular region of the thoracic cage in a sagittal plane.

The fifth rib is identified in the mid-axillary line. The following muscles are identified easily overlying the fifth rib: the latissimusdorsi (superficial and posterior),teres major (superior), and serratus muscle (deep and inferior).

As an extra-reference point, the thoracodorsal artery is used to aid the identification of the plane superficial to the serratus muscle. The needle (22G, 50-mm Tuohy needle) is introduced in-plane concerning the ultrasound Probe targeting the plane superficial to the serratus muscle.

Under continuous ultrasound guidance, a local anesthetic solution is injected then a catheter is threaded and Level of spread of analgesia in the SAPB group by cold and pinprick testing of the chest wall between T2 and T8/9 (assessed by an on-duty ICU resident who was unaware of the present study on the 1st postoperative day). Ultrasound-guided SAPB was done using a serratus anterior catheter Group DL (n=20) received a bolus of 30 mL of 0.25% bupivacaine followed by a continuous infusion of 0.125% bupivacaine at a rate of 7-12 ml/hr according to patient response upon ICU arrival after the stabilization of the clinical status. The infusion was continued until the end of the 1st 24 hours postoperatively .

GROUP 2: Thoracic epidural :

A thoracic epidural catheter was done to the patient while sitting. Tuohy needles are used. Epidural space can be identified by loss of resistance. Injection begins with a negative aspiration and a test dose (3 ccs of 1.5% lidocaine with 1:200,000 epinephrine) .A Continuous epidural technique through the placement of a catheter 3-5 cm beyond the needle is applied. Injection in 5ml increments of 0.25% bupivacaine is used until the block of the required segments achieved ( 10 to 15ml). sensory testing is via pinprick and cold test to detect sympathetic block . Throughout the technique hourly injection of 5 ml 0.25% bupivacaine for maintenance.

Both groups will have catheters covered by a sterile dressing and the area covered by the dressing will be extended to be the same for both groups. The anesthesiologist who will collect the data, and all the staff, other than the anesthesiologist inserting the catheter, are all blinded to the site of the catheter insertion . Catheter and infusion will be continued for 24 hours postoperatively.

Anaesthesia Management:

Inside OR ( operation room) The patient who is fasting for at least six hours before surgery and will be monitored continuously using electrocardiography, noninvasive blood pressure, peripheral oxygen saturation, and end-tidal carbon dioxide - using the Datex-Ohmeda S5 anesthesia monitor, model no: USE1913A - throughout the surgical procedure. Venous access and monitoring are installed before the regional technique.

Induction of general anesthesia will be performed for both groups using a regimen of IV fentanyl 2 μcg/kg, propofol 2 mg /kg, and rocuronium 0.5 mg/kg. Anesthesia will be maintained with inhaled sevoflurane with MAC 2-2.5% in oxygen;-enriched air (FiO2=50%) and top-up doses of rocuronium (0.1 mg/kg) IV will be administered by time every 45 minutes.

All patients will receive 1 g of IV paracetamol. Titrating doses of fentanyl (0.05-0.1 mic/kg) will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.

Ringer acetate will be infused to replace their fluid deficit, maintenance, and losses, and the patients will be mechanically ventilated at an appropriate setting that keeps end-tidal CO2 at 30-35mmHg.

One reading of mean arterial pressure and heart rate will be taken before induction of general anesthesia to be defined as a baseline reading and then will be recorded immediately before surgical incision and at 30 min intervals intraoperatively.

Hypotension (a decline of systolic blood pressure >20 % of the baseline) will be treated with 0.9% normal saline and/or 5mg ephedrine in incremental doses to maintain mean blood pressure above 70 mmHg.

The residual neuromuscular blockade will be reversed using Sugammadex (2 mg/kg), and extubation will be performed after complete recovery of the airway reflexes.

Extubated patients will be transferred to post-anesthesia care unit(PACU) where pain scores and MAP and heart rate will be recorded immediately on arrival and at 2, 4, 6, 12, and 24 h postoperatively in ICU and rescue analgesia will be provided in the form of morphine 3-5 mg I.V doses (according to the patient demand) In PACU (PACU discharge criteria: The modified Aldrete scoring system for determining when patients are ready for discharge from the postanesthesia care unit Discharge Criteria from Postanesthesia Care Unit Score Activity: able to move voluntarily or on command Four extremities 2 ,Two extremities 1, Zero extremities 0 and Respiration: Able to breathe deeply and cough freely 2, Dyspnea, shallow or limited breathing 1, Apneic 0 and Circulation: Blood pressure 20 mm of preanesthesia level 2, Blood pressure 20-50 mm preanesthesia level 1 ,Blood pressure 50 mm of preanesthesia level 0 and Consciousness :Fully awake 2 ,Arousable on calling 1, Not responding 0 and O2 saturation: Able to maintain O2 saturation >92% on room air 2, Needs O2 inhalation to maintain O2 saturation >90% 1 , O2 saturation <90% even with O2 supplementation 0) A score≥9 was required for discharge. ) . The total amount of morphine given in 24 h will be recorded in the two groups. Side effects such as nausea, vomiting, hypotension, bradycardia, over sedation will be recorded.

Postoperative nausea and vomiting (PONV) will be rated on a four-point verbal scale (none =no nausea, mild =nausea but no vomiting, moderate =vomiting one attack, severe =vomiting >one attack). 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting.

Sedation will be assessed in the recovery room with Ramsay scores (1 = anxious or restless or both; 2 = cooperative, orientated, and tranquil; 3 = responding to commands; 4 = brisk response to a stimulus; 5 = sluggish response to a stimulus, and 6 = no response to stimulus) excessively high sedation levels with Ramsay 5 or 6; adequate sedation levels needing observation with Ramsay 2 to 4; inadequate or insufficient sedation levels with Ramsay 1.

All Patients in our study will be transferred to ICU where the same recording protocol continues .

Statistical Analysis

The collected data will be, tabulated, and statistically analyzed using SPSS program (Statistical Package for Social Sciences) software version 20.0 Descriptive statistics were done for numerical parametric data as mean±SD (standard deviation) and minimum & maximum of the range and for numerical non parametric data as median and 1st& 3rd inter-quartile range, while they were done for categorical data as number and percentage.

Inferential analyses were done for quantitative variables using independent t-test in cases of two independent groups with parametric data and Mann Whitney U in cases of two independent groups with non parametric data.

Inferential analyses were done for qualitative data using Chi square test for independent groups. The level of significance was taken at P value <0.050 is significant, otherwise is non significant. The p-value is a statistical measure for the probability that the results observed in a study could have occurred by chance.

Sample size Using power and sample size calculator for intervention study ; with 0.05 alpha error and power of the study 0.80 and -0.5 non inferiority margin to calculate minimal sample size needed to Efficacy of perioperative US guided Serratus anterior plane block versus Thoracic epidural in adult patient undergoing Thoracotomy

* According to literature total 24 hrs' morphine consumption by group SAPB was 10.3±3 mg/24h. While it was 9.6± 4.3 mg/24 for group TEA The sample size calculated is 74 persons (37 in each arm of the study)

Sampling technique:

A convenient sample of patients with the inclusion and exclusion criteria will be assigned to the study. Each patient will be randomly allocated to each arm of the study using concealed random allocation technique till reaching total sample size calculated

ELIGIBILITY:
Inclusion Criteria:

* Physical status ASA II and III.
* Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.
* A patient undergoing thoracotomy for cancer surgery (Lobectomy, Pneumonectomy, and Decortication).

Exclusion Criteria:

* Patient refusal
* Known sensitivity or contraindication to local anesthetics.
* History of psychological disorders.
* Localized infection at the site of block.
* Coagulopathies with a platelet count below 50,000 or an INR>1.5: hereditary (e.g. hemophilia, fibrinogen abnormalities & deficiency of factor II) - acquired (e.g. impaired liver functions with PC less than 60 %, vitamin K deficiency &therapeutic anticoagulants drugs),History of unexplained or easy bruising and Prolonged bleeding from small cuts or after dental procedures.
* patients need prolonged mechanical ventilation postoperatively excluded from our study.
* failed blocks will be excluded from our study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative total morphine requirement. | 24 hours
  Postoperative total morphine requirement.

SECONDARY OUTCOMES:
Intraoperative fentanyl requirement. | 300 minutes
  Intraoperative fentanyl requirement.
Time to the first analgesia requested by the patient. | 24 hours
  time from postoperative period until the patinets asks for analgesia
Postoperative pain | 24 hours
  pain scores according to VAS score
Length of hospital stay. | 2 weeks
  time until discharge from the hospital
Patient satisfactory score | 24 hours
  patients will be classified either satisfied or not

CONTACTS AND LOCATIONS:
Overall Officials: Ashgan R Ali, Professor, Study Chair — Anaesthesiology Faculty of Medicine - Cairo University; Heba I Ahmed, Ass. Professor, Study Director — Anaesthesiology Faculty of Medicine - Cairo University; Reham M Gamal, Lecturer, Study Director — Anaesthesiology National Cancer Institute - Cairo University; Sylvia Samy Bassily Morgan, Master, Principal Investigator — Anaesthesiology National Cancer Institute - Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt